CLINICAL TRIAL: NCT02465515
Title: A Long Term, Randomised, Double Blind, Placebo-controlled Study to Determine the Effect of Albiglutide, When Added to Standard Blood Glucose Lowering Therapies, on Major Cardiovascular Events in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Albiglutide, When Added to Standard Blood Glucose Lowering Therapies, on Major Cardiovascular Events in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116174; 2014-001824-32 (EudraCT Number)
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: cardiovascular events /outcomes; Type 2 diabetes mellitus; albiglutide; glucagon-like peptide-1 receptor agonist
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albiglutide (Experimental): Albiglutide once weekly by subcutaneous injection. Starting dose 30 mg may be increased to 50 mg if needed. Albiglutide will be administered in addition to standard therapy for diabetes and cardiovascular health.
  Interventions: Biological: Albiglutide 30 mg; Biological: Albiglutide 50 mg
- Placebo (Placebo Comparator): Placebo once weekly by subcutaneous injection. Placebo will be administered in addition to standard therapy for diabetes and cardiovascular health.
  Interventions: Biological: Albiglutide matching placebo

INTERVENTIONS:
Biological: Albiglutide 30 mg — Once weekly subcutaneous injection. Starting dose 30 mg may be increased to 50 mg if needed.
  Arms: Albiglutide
Biological: Albiglutide 50 mg — Once weekly subcutaneous injection. Starting dose 30 mg may be increased to 50 mg if needed.
  Arms: Albiglutide
Biological: Albiglutide matching placebo — Once weekly subcutaneous injection. Matched to 30 mg and 50 mg albiglutide.
  Arms: Placebo

SUMMARY:
Albiglutide is an analogue of glucagon-like peptide-1 (GLP-1), used to treat type 2 diabetes This study will test whether albiglutide affects the occurrence of major cardiovascular events such as heart attacks or strokes and other important medical outcomes in persons with type 2 diabetes, when used alone or added to other diabetes treatments.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 40 years old. Women must be post-menopausal or using a highly effective method for avoidance of pregnancy.
* Diagnosis of type 2 diabetes.
* Established cardiovascular disease with at least one of the following: coronary artery disease, cerebrovascular disease, or peripheral arterial disease.
* HbA1c >7.0% (53 mmol/mol) (based on the most recent documented laboratory measurement within 6 months).
* Able and willing to provide informed consent.

Exclusion Criteria:

* Severely reduced kidney function: eGFR <30 ml/min/1.73 m^2 (based on the last measured and documented laboratory measurement within 6 months) or renal replacement therapy.
* Use of a GLP-1 receptor agonist at Screening.
* Severe gastroparesis
* History of pancreatitis or considered clinically at significant risk of developing pancreatitis during the course of the study.
* Personal or family history of medullary carcinoma of the thyroid or subject with multiple endocrine neoplasia type 2 (MEN-2). Personal history of pancreatic neuroendocrine tumours.
* Medical history which might limit the subject's ability to take trial treatments for the duration of the study or to otherwise complete the study.
* Breastfeeding, pregnancy, or planning a pregnancy during the course of the study. Note: a pregnancy test will be performed on all women of child bearing potential prior to study entry.
* Known allergy to any GLP-1 receptor agonist or excipients of albiglutide.
* Use of another investigational product within 30 days or according to local regulations, or currently enrolled in a study of an investigational device.
* Any other reason the investigator deems the subject to be unsuitable for the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9463 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (473):
- United States (128):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Goodyear, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Lancaster, California
  - GSK Investigational Site, Lomita, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Moreno Valley, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Marino, California
  - GSK Investigational Site, San Ramon, California
  - GSK Investigational Site, Simi Valley, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Belle Glade, Florida
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Fleming Island, Florida
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Lakeland, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Ponte Vedra, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Conyers, Georgia
  - GSK Investigational Site, Cumming, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Dunwoody, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Champaign, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, Moline, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Franklin, Indiana
  - GSK Investigational Site, Greenfield, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Munster, Indiana
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Lewiston, Maine
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Saint Cloud, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Rocky Mount, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Sandusky, Ohio
  - GSK Investigational Site, Springfield, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Feasterville, Pennsylvania
  - GSK Investigational Site, Harleysville, Pennsylvania
  - GSK Investigational Site, Jersey Shore, Pennsylvania
  - GSK Investigational Site, Lansdale, Pennsylvania
  - GSK Investigational Site, Newport, Pennsylvania
  - GSK Investigational Site, Penndel, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Pawtucket, Rhode Island
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Myrtle Beach, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Huntsville, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Suite 101, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Federal Way, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Madison, Wisconsin
- Argentina (16):
  - GSK Investigational Site, Adrogué, Buenos Aires
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Pergamino, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Godoy Cruz, Mendoza Province
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Berazategui
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Santa Fe
- Belgium (6):
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
- Bulgaria (6):
  - GSK Investigational Site, Byala
  - GSK Investigational Site, Gabrovo
  - GSK Investigational Site, Montana
  - GSK Investigational Site, Sevlievo
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
- Canada (29):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Cambridge, Ontario
  - GSK Investigational Site, Cornwall, Ontario
  - GSK Investigational Site, Corunna, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Smiths Falls, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Brossard, Quebec
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Lévis, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Saint-Lambert, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (9):
  - GSK Investigational Site, Beroun
  - GSK Investigational Site, Krnov
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Příbram
  - GSK Investigational Site, Uherské Hradiště
  - GSK Investigational Site, Ústí nad Labem
  - GSK Investigational Site, Zlín
- Denmark (10):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Esbjerg
  - GSK Investigational Site, Frederikssund
  - GSK Investigational Site, Hellerup
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Holbæk
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, København NV
  - GSK Investigational Site, København S
  - GSK Investigational Site, Roskilde
- France (11):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Broglie
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Narbonne
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (50):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Ludwigsburg, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Elsterwerda, Brandenburg
  - GSK Investigational Site, Falkensee, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Stuhr, Lower Saxony
  - GSK Investigational Site, Wardenburg, Lower Saxony
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Kleve, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Bad Kreuznach, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Sankt Ingbert, Saarland
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Oschatz, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Riesa, Saxony
  - GSK Investigational Site, Schkeuditz, Saxony
  - GSK Investigational Site, Hohenmölsen, Saxony-Anhalt
  - GSK Investigational Site, Jerichow, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Dortmund
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Mannheim
  - GSK Investigational Site, München
- Greece (9):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Lamia
  - GSK Investigational Site, Nikaia Piraeus
  - GSK Investigational Site, Piraeus
  - GSK Investigational Site, Thessaloniki
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin
- Hungary (9):
  - GSK Investigational Site, Baja
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Eger
  - GSK Investigational Site, Gödöllő
  - GSK Investigational Site, Hatvan
  - GSK Investigational Site, Komárom
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Sátoraljaújhely
- Italy (19):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, San Giovanni Rotondo (FG), Apulia
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Arenzano (GE), Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Vigevano (PV), Lombardy
  - GSK Investigational Site, Olbia (OT), Sardinia
  - GSK Investigational Site, Ancona, The Marches
  - GSK Investigational Site, Ascoli Piceno, The Marches
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, S.Andrea Delle Fratte - S. Sisto (PG), Umbria
  - GSK Investigational Site, Padua, Veneto
- Mexico (10):
  - GSK Investigational Site, Aguascalientes, Ags, Aguascalientes
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Tlaquepaque, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Monterrey NL, Nuevo León
  - GSK Investigational Site, Querétaro City, Querétaro
  - GSK Investigational Site, Mazatlán, Sinaloa
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, Mexico City
- Netherlands (10):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Gouda
  - GSK Investigational Site, Hardenberg
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hoogeveen
  - GSK Investigational Site, Meppel
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sneek
- Norway (4):
  - GSK Investigational Site, Hoenefoss
  - GSK Investigational Site, Kolbjørnsvik
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
- Peru (6):
  - GSK Investigational Site, Trujillo, La Libertad
  - GSK Investigational Site, San Martín de Porres, Lima region
  - GSK Investigational Site, Callao, Lima
  - GSK Investigational Site, Arequipa
  - GSK Investigational Site, Lima
  - GSK Investigational Site, Piura
- Philippines (3):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Laoag
- Poland (12):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gniewkowo
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wierzchosławice
  - GSK Investigational Site, Wroclaw
- Russia (19):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- South Africa (9):
  - GSK Investigational Site, Bloemfontein, Free State
  - GSK Investigational Site, Tongaat, KwaZulu-Natal
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Houghton Estate
  - GSK Investigational Site, Kuilsrivier
  - GSK Investigational Site, Paarl
  - GSK Investigational Site, Pinelands
  - GSK Investigational Site, Umhlanga
- South Korea (8):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Gyeonggido
  - GSK Investigational Site, Kangwondo
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
  - GSK Investigational Site, Suwon, Kyonggi-do
- Spain (29):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Alzira/Valencia
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Badalona / Barcelona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Boadilla Del Monte (Madrid)
  - GSK Investigational Site, Canet de Mar - Barcelona
  - GSK Investigational Site, Cangas Del Narcea/Asturias
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Granada
  - GSK Investigational Site, León
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Sagunto/Valencia
  - GSK Investigational Site, San Juan (Alicante)
  - GSK Investigational Site, Sanlucar de Barrameda - Cádiz
  - GSK Investigational Site, Santa Coloma de Gramanet (Barcelona)
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Tarrasa, Barcelona
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo-Pontevedra
- Sweden (15):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Eksjö
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Härnösand
  - GSK Investigational Site, Helsingborg
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Kristianstad
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Ljungby
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Rättvik
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Uppsala
- Taiwan (6):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Hualien City
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- Thailand (4):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Pathum Thani
  - GSK Investigational Site, Songkhla
- Ukraine (11):
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kherson
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolaiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Uzhhorod
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhya
- United Kingdom (23):
  - GSK Investigational Site, Soham, Cambridgeshire
  - GSK Investigational Site, Chesterfield, Derbyshire
  - GSK Investigational Site, Romford, Essex
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Trowbridge, Wiltshire
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, Axbridge, Somerset
  - GSK Investigational Site, Ayr
  - GSK Investigational Site, Blackpool
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Dumfries
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Fife
  - GSK Investigational Site, Gloucester
  - GSK Investigational Site, Lancaster
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newport
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Rotherham
  - GSK Investigational Site, Sidcup, Kent
  - GSK Investigational Site, Trowbridge
  - GSK Investigational Site, Wigan

REFERENCES:
- [Background] John McMurray, Stefano Del Prato, Adrian Hernandez, Larry Leiter, Chris Granger, Ralph D'Agostino, Jennifer Green, Kristina Sigmon, Anne Rosenberg Nigel Jones, Karl Thorpe, Matt Somerville, Salim Janmohamed. Albiglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes and Cardiovascular Disease. Lancet. 2018
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Gilbert MP, Skelly J, Hernandez AF, Green JB, Krychtiuk KA, Granger CB, Leiter LA, McMurray JJV, Del Prato S, Pratley RE. Effect of albiglutide on cardiovascular outcomes in older adults: A post hoc analysis of a randomized controlled trial. Diabetes Obes Metab. 2024 May;26(5):1714-1722. doi: 10.1111/dom.15479. Epub 2024 Feb 6. PMID 38317618
- [Derived] O'Brien EC, Raman SR, Ellis A, Hammill BG, Berdan LG, Rorick T, Janmohamed S, Lampron Z, Hernandez AF, Curtis LH. The use of electronic health records for recruitment in clinical trials: a mixed methods analysis of the Harmony Outcomes Electronic Health Record Ancillary Study. Trials. 2021 Jul 19;22(1):465. doi: 10.1186/s13063-021-05397-0. PMID 34281607
- [Derived] Hernandez AF, Green JB, Janmohamed S, D'Agostino RB Sr, Granger CB, Jones NP, Leiter LA, Rosenberg AE, Sigmon KN, Somerville MC, Thorpe KM, McMurray JJV, Del Prato S; Harmony Outcomes committees and investigators. Albiglutide and cardiovascular outcomes in patients with type 2 diabetes and cardiovascular disease (Harmony Outcomes): a double-blind, randomised placebo-controlled trial. Lancet. 2018 Oct 27;392(10157):1519-1529. doi: 10.1016/S0140-6736(18)32261-X. Epub 2018 Oct 2. PMID 30291013
- [Derived] Green JB, Hernandez AF, D'Agostino RB, Granger CB, Janmohamed S, Jones NP, Leiter LA, Noronha D, Russell R, Sigmon K, Del Prato S, McMurray JJV. Harmony Outcomes: A randomized, double-blind, placebo-controlled trial of the effect of albiglutide on major cardiovascular events in patients with type 2 diabetes mellitus-Rationale, design, and baseline characteristics. Am Heart J. 2018 Sep;203:30-38. doi: 10.1016/j.ahj.2018.03.030. Epub 2018 Jun 12. PMID 30015066
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Generalizability of glucagon-like peptide-1 receptor agonist cardiovascular outcome trials enrollment criteria to the US type 2 diabetes population. Am J Manag Care. 2018 Apr;24(8 Suppl):S146-S155. PMID 29693361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, parallel group, placebo-controlled study in participants with Type 2 diabetes having a previous history of cardiovascular disease and not having optimal glycemic control.
Pre-assignment Details: A total of 10793 participants were screened of which 1330 failed screening and 9463 participants were randomized in a 1:1 ratio to receive either once weekly albiglutide or matching placebo subcutaneous injections. The study was conducted in 28 countries
Groups:
- Placebo: Albiglutide matching placebo was administered once weekly as subcutaneous injection in the abdomen, thigh or upper arm region in addition to the standard of care therapy for diabetes and cardiovascular health.
- Albiglutide: Albiglutide was administered once weekly as subcutaneous injection in the abdomen, thigh or upper arm region. Participants were administered albiglutide at a dose of 30 milligrams (mg) or 50 mg once weekly in addition to the standard of care therapy for diabetes and cardiovascular health.
Period: Overall Study
Arm/Group | Placebo | Albiglutide
Started | 4732 | 4731
Completed | 4578 | 4620
Not Completed | 154 | 111
Not completed — Investigator site closed | 4 | 5
Not completed — Withdrawal by Subject | 74 | 43
Not completed — Physician Decision | 8 | 12
Not completed — Lost to Follow-up | 68 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Albiglutide | Total
Number analyzed (Participants) | 4732 | 4731 | 9463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.65) | 64.1 (8.71) | 64.1 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1467 | 1427 | 2894
  Male | 3265 | 3304 | 6569
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, customized: American Indian (Amer. Ind.) or Alaska Native | 238 | 280 | 518
  Race, customized: Central/South Asian Heritage (Her.) | 27 | 25 | 52
  Race, customized: Japanese Her./East Asian Her/South East Asian Her. | 215 | 204 | 419
  Race, customized: Black or African American (Amer.) | 118 | 121 | 239
  Race, customized: Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Race, customized: White | 4024 | 4006 | 8030
  Race, customized: Amer Ind. or Alaska Native & Black or African Amer | 1 | 3 | 4
  Race, customized: Asian & Black or African Amer. | 1 | 0 | 1
  Race, customized: Asian & White | 0 | 1 | 1
  Race, customized: Black or African Amer. & White | 81 | 67 | 148
  Race, customized: Unknown | 1 | 1 | 2
  Race, customized: Amer. Ind. or Alaska Native & White | 24 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Major Adverse Cardiovascular Events (MACE) During Cardiovascular (CV) Follow-up Time Period
Description: Time to MACE defined as the time to first occurrence of Cardiovascular Endpoint Committee (CEC)-adjudicated MACE (CV death, myocardial infarction [MI] or stroke) was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period. The analysis was performed on the Intent to Treat (ITT) Population which comprised of all randomized participants excluding participants who did not provide consent.
Time Frame: Median of 1.65 person years for CV follow-up time period
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Events per 100 person years | 5.87 [5.33 to 6.45] | 4.57 [4.10 to 5.08]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Non-Inferiority — Non-inferiority was determined by testing the hypothesis that the observed hazard ratio is significantly different from the null margin of 1.3 (a one-sided p <0.025 for such a test with result in appropriate direction being equivalent to the upper 95% confidence limit for the hazard ratio being less than 1.3); p < 0.0001, Wald test — One-sided p-value based on Wald test of hazard ratio (HR) >=1.3 versus HR <1.3; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.68 to 0.90] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate
Statistical Analysis 2: Comparison: Placebo vs Albiglutide; Test type: Superiority; p < 0.001, Wald test — Two-sided p-value based on Wald test of HR=1 versus HR not equal to 1

2. Secondary Outcome: Time to First Occurrence of MACE or Urgent Revascularization for Unstable Angina
Description: Time to first occurrence of CEC-adjudicated MACE (CV death, MI or stroke) or urgent revascularization for unstable angina was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Median of 1.65 person years for CV follow-up time period
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Events per 100 person years | 6.45 [5.88 to 7.06] | 5.06 [4.56 to 5.60]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, Wald statistic — Two-sided p-value based on the Wald statistic; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.69 to 0.90] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

3. Secondary Outcome: Time to Adjudicated CV Death
Description: Time to adjudicated CV death was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Median of 1.65 person years for the CV follow-up time period
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Events per 100 person years | 1.72 [1.44 to 2.04] | 1.61 [1.33 to 1.92]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p = 0.578, Wald statistic — Two-sided p-value based on the Wald statistic; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.73 to 1.19] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

4. Secondary Outcome: Time to First Occurrence of Adjudicated MI
Description: Time to first occurrence of adjudicated MI was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Median of 1.65 person years for CV follow-up time period
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Events per 100 person years | 3.26 [2.86 to 3.70] | 2.43 [2.09 to 2.81]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p = 0.003, Wald statistic — Two-sided p-value based on the Wald statistic; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.61 to 0.90] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

5. Secondary Outcome: Time to First Occurrence of Adjudicated Stroke
Description: Time to first occurrence of adjudicated stroke was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Median of 1.65 person years for CV follow-up time period
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Events per 100 person years | 1.45 [1.19 to 1.74] | 1.25 [1.01 to 1.53]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p = 0.300, Wald statistic — Two-sided p-value based on the Wald statistic; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.66 to 1.14] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

6. Secondary Outcome: Time to First Occurrence of Adjudicated CV Death or Hospitalization for Heart Failure (HF)
Description: Time to first occurrence of adjudicated CV death or hospitalization for HF was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Median of 1.65 person years for CV follow-up time period
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Events per 100 person years | 2.92 [2.55 to 3.34] | 2.49 [2.15 to 2.88]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p = 0.113, Wald statistic — Two-sided p-value based on the Wald statistic; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.70 to 1.04] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

7. Secondary Outcome: Time to Initiation of Insulin of More Than 3 Months Duration for Those Participants Not Treated With Insulin at Study Start
Description: Time to initiation of insulin of more than 3 months duration in participants not treated with insulin at study start was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the on-therapy and post-therapy AE time period. The analysis was performed on Non-Insulin Population which comprised of participants in the ITT Population who were not on insulin at Baseline.
Time Frame: Up to 2.7 years
Population: Non-Insulin Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 1995 | 1871
Events per 100 person years | 8.58 [7.56 to 9.70] | 3.56 [2.92 to 4.31]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Superiority; p < 0.001, Wald test — Two-sided p-value based on Wald test of HR=1 versus HR not equal to 1; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.33 to 0.53] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

8. Secondary Outcome: Time to Initiation of Prandial Insulin in Those Participants on Basal Insulin at Study Start
Description: Time to initiation of prandial insulin in those participants on basal insulin at study start was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the on-therapy and post-therapy AE time period. The analysis was performed on Basal Insulin Population which comprised of participants in the ITT Population who were on basal insulin but not on other insulin at Baseline (i.e., will not include a participant on a mixed insulin or on a prandial-only insulin).
Time Frame: Up to 2.7 years
Population: Basal Insulin Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 1040 | 1028
Events per 100 person years | 5.09 [4.06 to 6.31] | 3.59 [2.73 to 4.63]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Superiority; p = 0.043, Wald test — Two-sided p-value based on Wald test of HR=1 versus HR not equal to 1; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.51 to 0.99] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

9. Secondary Outcome: Percentage of Participants Achieving Composite Metabolic Endpoint
Description: Percentage of participants achieving composite metabolic endpoint defined as the percentage of participants achieving glycemic control (glycated hemoglobin [HbA1c] <=7% ) with no severe hypoglycemic incidents and weight gain < 5%. Final Assessment is the latest post-Baseline assessment of both HbA1c and weight.
Time Frame: Months 8, 16, 24 and final assessment (up to 2.7 years)
Population: ITT Population. Only those participants with HbA1c and weight values at Baseline and at the specified visits were analyzed (represented by n=X in category titles)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Percentage of participants
  Month 8, n=4127, 4195: number analyzed (Participants) | 4127 | 4195
  Month 8, n=4127, 4195 | 15.4 | 32.2
  Month 16, n=3026, 3118: number analyzed (Participants) | 3026 | 3118
  Month 16, n=3026, 3118 | 16.5 | 28.7
  Month 24, n=1119, 1173: number analyzed (Participants) | 1119 | 1173
  Month 24, n=1119, 1173 | 17.8 | 28.6
  Final assessment, n=4401, 4455: number analyzed (Participants) | 4401 | 4455
  Final assessment, n=4401, 4455 | 15.1 | 26.0
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, Mantel Haenszel — P-value based on the covariate-adjusted extended Mantel-Haenszel test. Covariates include Baseline HbA1c (<8.0% versus >= 8.0%) and Baseline diabetes therapy (diet and exercise alone versus all other therapies); Month 8
Statistical Analysis 2: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, Mantel Haenszel — [p-value comment as in outcome 9, analysis 1]; Month 16
Statistical Analysis 3: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, Mantel Haenszel — [p-value comment as in outcome 9, analysis 1]; Month 24
Statistical Analysis 4: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, Mantel Haenszel — [p-value comment as in outcome 9, analysis 1]; Final assessment

10. Secondary Outcome: Time to First Occurrence of a Clinically Important Microvascular Event
Description: Clinically important microvascular events were defined as the following: need for renal transplant or dialysis, new diabetes-related blindness, and procedures (laser photocoagulation or anti-vascular endothelial growth factor treatment or vitrectomy for diabetic retinopathy/eye disease). Time to first occurrence of a clinically important microvascular event was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% confidence interval. First event person-years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the on-therapy and post-therapy AE time period.
Time Frame: Up to 2.7 years
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Events per 100 person years | 0.69 [0.52 to 0.90] | 0.46 [0.32 to 0.63]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Superiority; p = 0.055, Wald test — Two-sided p-value based on Wald test of HR=1 versus HR not equal to 1; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.43 to 1.01] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

11. Secondary Outcome: Change From Baseline in HbA1c
Description: Change from Baseline in HbA1c was analyzed using mixed model repeated measures (MMRM) including observed case data (does not impute any missing data). Baseline is the last non-missing value assessed on or before treatment start date. Change from Baseline is the value at specified time point minus the Baseline value. Change from Baseline in HbA1c using Baseline data from Local or Central Laboratory, and post-Baseline Central Laboratory data is presented.
Time Frame: Baseline and Months 8 and 16
Population: ITT Population. Only those participants with value at Baseline and at the specified visit is presented (represented by n=X in category titles)
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Percentage of HbA1c
  Month 8, n=4211, 4289: number analyzed (Participants) | 4211 | 4289
  Month 8, n=4211, 4289 | -0.28 (0.020) | -0.92 (0.019)
  Month 16, n=3066, 3163: number analyzed (Participants) | 3066 | 3163
  Month 16, n=3066, 3163 | -0.31 (0.023) | -0.83 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, t-test, 2 sided — P-value from a two-sided t-test to test whether the difference of least square means (Albiglutide - Placebo) is equal to zero; Mean Difference (Net) = -0.63, 95% CI 2-sided [-0.69 to -0.58] — Based on MMRM model: Change=Baseline HbA1c+Treatment+Visit+Treatment-by-Visit Interaction+Baseline HbA1c-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 8
Statistical Analysis 2: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -0.52, 95% CI 2-sided [-0.58 to -0.45] — Based on MMRM model: Change=Baseline HbA1c+Treatment+Visit+Treatment-by-Visit Interaction+Baseline HbA1c-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 16

12. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from Baseline in body weight was analyzed using mixed model repeated measures including observed case data (does not impute any missing data). Baseline is the last non-missing value assessed on or before treatment start date. Change from Baseline is the value at specified time point minus the Baseline value.
Time Frame: Baseline and Months 8 and 16
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Kilograms
  Month 8, n=4217, 4286: number analyzed (Participants) | 4217 | 4286
  Month 8, n=4217, 4286 | -0.36 (0.062) | -1.02 (0.061)
  Month 16, n=3068, 3173: number analyzed (Participants) | 3068 | 3173
  Month 16, n=3068, 3173 | -0.53 (0.084) | -1.36 (0.083)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, t-test, 2 sided — P-value from a two-sided t-test to test whether the difference of least square means (Albiglutide-Placebo) is equal to zero; Mean Difference (Net) = -0.66, 95% CI 2-sided [-0.83 to -0.49] — Based on MMRM model: Change=Baseline Body Weight+Treatment+Visit+Treatment-by-Visit Interaction+Baseline Body Weight-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 8
Statistical Analysis 2: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = -0.83, 95% CI 2-sided [-1.06 to -0.60] — Based on MMRM model: Change=Baseline Body Weight+Treatment+Visit+Treatment-by-Visit Interaction+Baseline Body weight-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 16

13. Secondary Outcome: Change From Baseline in Treatment Related Impact Measures-Diabetes (TRIM-D) Total Score
Description: The TRIM-D is a 28 item treatment satisfaction measure with 5 domains assessing Treatment Burden, Daily Life, Diabetes Management, Compliance and Psychological Health. The raw score ranges for each subscale were: treatment burden (6 to 30), daily life (5 to 25), diabetes management (5 to 25), compliance (4 to 20) and psychological health (8 to 40), higher scores indicating better health state. Total raw score was determined by summing the raw scores for each of the subscales and the total score (transformed) was determined as [(raw score minus lowest possible raw score)/possible raw score range] x100. The possible total (transformed) score range is 0-100, where higher scores indicated better health state. Baseline is the last non-missing value assessed on or before treatment start date. Change from Baseline is the value at specified time point minus the Baseline value.
Time Frame: Baseline and Months 8 and 16
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Scores on a scale
  Month 8, n=3013, 3041: number analyzed (Participants) | 3013 | 3041
  Month 8, n=3013, 3041 | 4.53 (0.194) | 6.92 (0.193)
  Month 16, n=1738, 1840: number analyzed (Participants) | 1738 | 1840
  Month 16, n=1738, 1840 | 4.80 (0.247) | 7.13 (0.241)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = 2.39, 95% CI 2-sided [1.85 to 2.93] — Based on MMRM model: Change=Baseline Total Score+Treatment+Visit+Treatment-by-Visit Interaction+Baseline Total Score-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 8
Statistical Analysis 2: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = 2.33, 95% CI 2-sided [1.66 to 3.01] — Based on MMRM model: Change=Baseline Total Score+Treatment+Visit+Treatment-by-Visit Interaction+Baseline Total Score-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 16

14. Secondary Outcome: Change From Baseline in EuroQol- 5 Dimension (EQ-5D) Visual Analogue Scale (VAS) Score
Description: The EQ-5D is a standardized instrument used to evaluate generic health-related quality of life, comprising 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It provides a simple descriptive profile and a single index value for health status. The EQ-5D self-reported questionnaire includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. Baseline is the last non-missing value assessed on or before treatment start date. Change from Baseline is the value at specified time point minus the Baseline value.
Time Frame: Baseline and Months 8 and 16
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Scores on a scale
  Month 8, n=3982, 4014: number analyzed (Participants) | 3982 | 4014
  Month 8, n=3982, 4014 | 1.36 (0.217) | 2.83 (0.216)
  Month 16, n=2347, 2481: number analyzed (Participants) | 2347 | 2481
  Month 16, n=2347, 2481 | 1.87 (0.287) | 2.39 (0.279)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = 1.47, 95% CI 2-sided [0.87 to 2.07] — Based on MMRM model: Change=Baseline Score+Treatment+Visit+Treatment-by-Visit Interaction+Baseline Score-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 8
Statistical Analysis 2: Comparison: Placebo vs Albiglutide; Test type: Other; p = 0.192, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Mean Difference (Net) = 0.52, 95% CI 2-sided [-0.26 to 1.31] — Based on MMRM model: Change=Baseline Score+Treatment+Visit+Treatment-by-Visit Interaction+Baseline Score-by-Visit Interaction. Difference of least squares means (Albiglutide - Placebo) is from MMRM model for Month 16

15. Secondary Outcome: Time to Death
Description: Time to death was analyzed using a Cox Proportional Hazards regression model with treatment group as the only covariate. The incidence rate per 100 person years (100*number of participants who died/endpoint person-years) is presented along with 95% confidence interval. Endpoint person-years=(cumulative total time to event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the Vital Status follow-up time period.
Time Frame: Median of 1.73 years for the Vital Status follow-up time period
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4732 | 4731
Events per 100 person years | 2.56 [2.22 to 2.93] | 2.44 [2.11 to 2.81]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p = 0.644, Wald test — Two-sided p-value based on Wald test of HR=1 versus HR not equal to 1; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.79 to 1.16] — Hazard ratio is estimated using a Cox proportional hazard regression model with treatment as the only covariate

16. Secondary Outcome: Number of Participants With Non-fatal Serious Adverse Events (SAEs)
Description: SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before; is associated with liver injury and impaired liver function. Number of participants with on-therapy non-fatal SAEs are presented. Safety Population comprised of all randomized participants who received at least one dose of study treatment.
Time Frame: Up to 2.7 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4715 | 4717
Participants | 974 | 891

17. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation of Investigational Product (AELD)
Description: The number of participants with on-therapy AEs leading to discontinuation of investigational product is reported.
Time Frame: Up to 2.7 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4715 | 4717
Participants | 334 | 427

18. Secondary Outcome: Number of Participants With AEs of Special Interest
Description: The protocol defined AEs of special interest included: development of thyroid cancer; hematologic malignancy; pancreatic cancer; pancreatitis (investigator reported and pancreatitis positively adjudicated by the Pancreatic Adjudication Committee [PAC]); investigational product injection site reactions; immunological reactions; severe hypoglycemic events; hepatic events; hepatic enzyme elevations (including gamma glutamyl transferase [GGT]); serious gastrointestinal (GI) events; appendicitis; atrial fibrillation/flutter; pneumonia; worsening renal function and diabetic retinopathy. The number of participants with on-therapy AEs of special interest is reported.
Time Frame: Up to 2.7 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4715 | 4717
Participants
  Thyroid cancer diagnosis | 0 | 0
  Hematologic malignancy | 5 | 9
  Pancreatic cancer | 5 | 6
  Investigational product injection site reaction | 29 | 86
  Hypersensitivity | 48 | 45
  Severe hypoglycemic events | 55 | 31
  Hepatic events | 74 | 98
  Hepatic enzyme elevations (including GGT) | 34 | 51
  Serious GI Events | 87 | 92
  Appendicitis | 8 | 3
  Atrial fibrillation/atrial flutter | 131 | 108
  Pneumonia | 138 | 131
  Renal impairment | 319 | 279
  Diabetic retinopathy | 89 | 78
  Investigator-reported pancreatitis | 13 | 14
  Pancreatitis positively adjudicated by PAC | 7 | 10

19. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) Calculated Using Modification of Diet in Renal Disease (MDRD) Formula
Description: Blood samples were collected for the measurement of serum creatinine. Serum creatinine values were used to calculate eGFR using the MDRD formula, eGFR=175 x (serum creatinine)^-1.154 x (Age)^-0.203 x (0.742 if female) x (1.212 if African American). Baseline is the last non-missing value assessed on or before treatment start date. Change from Baseline is the value at specified time point minus the Baseline value. Change from Baseline in eGFR using Baseline data from Local or Central Laboratory, and post-Baseline Central Laboratory data for the on-treatment time period is presented.
Time Frame: Baseline and Months 8 and 16
Population: Safety Population. Only those participants with a value at Baseline and specified visit were analyzed (represented by n=X in category titles)
Measure: Least Squares Mean (Standard Error); unit: Milliliter/minute/1.73 meter square
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4715 | 4717
Milliliter/minute/1.73 meter square
  Month 8; n=3977,4008: number analyzed (Participants) | 3977 | 4008
  Month 8; n=3977,4008 | 1.22 (0.264) | 0.10 (0.262)
  Month 16; n=2354,2496: number analyzed (Participants) | 2354 | 2496
  Month 16; n=2354,2496 | -0.90 (0.303) | -1.33 (0.296)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide; Test type: Other; p = 0.003, t-test, 2 sided — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -1.11, 95% CI 2-sided [-1.84 to -0.39] — Based on MMRM model: Change=Baseline eGFR+Treatment+Visit+Treatment-by-Visit Interaction+Baseline eGFR-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 8
Statistical Analysis 2: Comparison: Placebo vs Albiglutide; Test type: Other; p = 0.315, t-test, 2 sided — [p-value comment as in outcome 12, analysis 1]; Mean Difference (Net) = -0.43, 95% CI 2-sided [-1.26 to 0.41] — Based on MMRM model: Change=Baseline eGFR+Treatment+Visit+Treatment-by-Visit Interaction+Baseline eGFR-by-Visit Interaction. Difference of least squares means (Albiglutide-Placebo) is from MMRM model for Month 16

20. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were taken with the participant in a semi-recumbent or seated position after at least a 5-minute rest period. Baseline is the last non-missing value assessed on or before treatment start date. Change from Baseline is the value at specified time point minus the Baseline value.
Time Frame: Baseline and Months 8,16,24 and end of study (up to 2.7 years)
Population: Safety Population. Only those participants with a value at Baseline and specified visit were analyzed (represented n=X in category titles)
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4715 | 4717
Millimeter of mercury
  SBP, Month 8; n=4241, 4319: number analyzed (Participants) | 4241 | 4319
  SBP, Month 8; n=4241, 4319 | -0.5 (17.33) | -1.0 (16.80)
  SBP, Month 16; n=3082, 3187: number analyzed (Participants) | 3082 | 3187
  SBP, Month 16; n=3082, 3187 | -0.5 (17.45) | -0.9 (17.58)
  SBP, Month 24; n=1133, 1198: number analyzed (Participants) | 1133 | 1198
  SBP, Month 24; n=1133, 1198 | -0.9 (18.62) | -1.2 (17.51)
  SBP, End of study; n=3897, 4015: number analyzed (Participants) | 3897 | 4015
  SBP, End of study; n=3897, 4015 | 0.0 (17.68) | -0.4 (17.58)
  DBP, Month 8; n=4241, 4319: number analyzed (Participants) | 4241 | 4319
  DBP, Month 8; n=4241, 4319 | -0.5 (10.26) | -0.4 (10.12)
  DBP, Month 16; n=3082, 3187: number analyzed (Participants) | 3082 | 3187
  DBP, Month 16; n=3082, 3187 | -0.9 (10.74) | -0.5 (10.39)
  DBP, Month 24; n=1133, 1198: number analyzed (Participants) | 1133 | 1198
  DBP, Month 24; n=1133, 1198 | -1.1 (10.87) | -1.0 (10.29)
  DBP, End of study; n=3897, 4015: number analyzed (Participants) | 3897 | 4015
  DBP, End of study; n=3897, 4015 | -0.7 (10.66) | -0.6 (10.57)

21. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured with the participant in a semi-recumbent or seated position after at least a 5-minute rest period. Baseline is the last non-missing value assessed on or before treatment start date. Change from Baseline is the value at specified time point minus the Baseline value.
Time Frame: Baseline and Months 8, 16, 24 and end of study (up to 2.7 years)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Albiglutide
Number analyzed (Participants) | 4715 | 4717
Beats per minute
  Month 8; n=4239, 4312: number analyzed (Participants) | 4239 | 4312
  Month 8; n=4239, 4312 | 0.2 (9.99) | 1.6 (10.07)
  Month 16; n=3078, 3181: number analyzed (Participants) | 3078 | 3181
  Month 16; n=3078, 3181 | 0.3 (10.19) | 1.6 (10.16)
  Month 24; n=1131, 1195: number analyzed (Participants) | 1131 | 1195
  Month 24; n=1131, 1195 | 0.6 (10.84) | 1.7 (10.32)
  End of study; n=3892, 4005: number analyzed (Participants) | 3892 | 4005
  End of study; n=3892, 4005 | 0.8 (10.64) | 1.8 (10.50)

ADVERSE EVENTS:
Time Frame: On-therapy non-SAEs and SAEs were reported on or after treatment start date and within 56 days after treatment stop date (Up to 2.7 years)
Description: SAEs, non-SAELDs and non-SAEs of pre-specified interest were reported systematically in the Safety Population. Some investigators collected other non-SAEs for some participants (i.e. non-systematically). CV events referred for adjudication as study endpoints were not duplicate reported as AEs. Deaths were reported for ITT Population.
Arm/Group | Albiglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 196/4731 | 205/4732
Serious Adverse Events (participants affected / at risk) | 932/4717 | 1022/4715
Other Adverse Events (participants affected / at risk) | 0/4717 | 0/4715
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albiglutide (N=4717) | Placebo (N=4715)
Pneumonia (Infections and infestations) | 74 (79) | 77 (81)
Acute kidney injury (Renal and urinary disorders) | 42 (46) | 47 (52)
Atrial fibrillation (Cardiac disorders) | 45 (48) | 41 (47)
Peripheral arterial occlusive disease (Vascular disorders) | 33 (37) | 41 (48)
Angina pectoris (Cardiac disorders) | 37 (38) | 36 (39)
Coronary artery disease (Cardiac disorders) | 24 (24) | 31 (31)
Sepsis (Infections and infestations) | 23 (23) | 28 (29)
Urinary tract infection (Infections and infestations) | 26 (27) | 23 (27)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (16) | 30 (42)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 21 (33)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (12) | 30 (34)
Cellulitis (Infections and infestations) | 20 (22) | 20 (20)
Non-cardiac chest pain (General disorders) | 15 (19) | 22 (23)
Diabetic foot (Skin and subcutaneous tissue disorders) | 14 (16) | 22 (26)
Renal impairment (Renal and urinary disorders) | 17 (17) | 12 (13)
Syncope (Nervous system disorders) | 14 (17) | 13 (15)
Death (General disorders) | 10 (10) | 14 (14)
Hypertension (Vascular disorders) | 11 (12) | 12 (12)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (9) | 16 (16)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 14 (16)
Bronchitis (Infections and infestations) | 10 (10) | 11 (12)
Erysipelas (Infections and infestations) | 9 (9) | 12 (14)
Atrial flutter (Cardiac disorders) | 6 (6) | 14 (15)
Osteomyelitis (Infections and infestations) | 6 (6) | 14 (14)
Peripheral ischaemia (Vascular disorders) | 7 (11) | 13 (13)
Cholelithiasis (Hepatobiliary disorders) | 12 (12) | 7 (7)
Gangrene (Infections and infestations) | 6 (6) | 13 (14)
Hypertensive crisis (Vascular disorders) | 8 (8) | 11 (11)
Chest pain (General disorders) | 8 (8) | 10 (10)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (12) | 10 (10)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 10 (10)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 (4) | 13 (13)
Hypotension (Vascular disorders) | 10 (10) | 7 (7)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 12 (12)
Atrioventricular block complete (Cardiac disorders) | 11 (11) | 5 (5)
Carotid artery stenosis (Nervous system disorders) | 9 (11) | 7 (7)
Gastroenteritis (Infections and infestations) | 8 (8) | 8 (8)
Peripheral vascular disorder (Vascular disorders) | 3 (3) | 13 (19)
Renal failure (Renal and urinary disorders) | 9 (10) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (7)
Ventricular tachycardia (Cardiac disorders) | 6 (7) | 9 (10)
Cardiac failure (Cardiac disorders) | 10 (10) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 10 (11)
Urosepsis (Infections and infestations) | 6 (6) | 8 (8)
Cardiogenic shock (Cardiac disorders) | 9 (9) | 4 (4)
Diabetic foot infection (Infections and infestations) | 4 (6) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 7 (8) | 6 (7)
Gastritis (Gastrointestinal disorders) | 5 (5) | 8 (8)
Myocardial ischaemia (Cardiac disorders) | 6 (6) | 7 (7)
Bradycardia (Cardiac disorders) | 8 (8) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 9 (10)
Cataract (Eye disorders) | 7 (7) | 5 (6)
Cholecystitis (Hepatobiliary disorders) | 7 (7) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 9 (9)
Extremity necrosis (Vascular disorders) | 7 (7) | 5 (6)
Multiple organ dysfunction syndrome (General disorders) | 6 (6) | 6 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (9)
Cholecystitis acute (Hepatobiliary disorders) | 7 (7) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 9 (9) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 2 (2)
Septic shock (Infections and infestations) | 4 (4) | 7 (7)
Cardio-respiratory arrest (Cardiac disorders) | 5 (5) | 5 (6)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 8 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (6)
Orthostatic hypotension (Vascular disorders) | 4 (5) | 6 (6)
Postoperative wound infection (Infections and infestations) | 6 (6) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 5 (6)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Appendicitis (Infections and infestations) | 2 (2) | 7 (7)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (4) | 5 (5)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 6 (6)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Cardiac arrest (Cardiac disorders) | 4 (4) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 6 (7) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 4 (6) | 5 (6)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (5)
Aortic stenosis (Vascular disorders) | 4 (4) | 4 (4)
Asthenia (General disorders) | 4 (4) | 4 (4)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 7 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Haematuria (Renal and urinary disorders) | 5 (5) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 5 (5)
Inguinal hernia (Gastrointestinal disorders) | 6 (6) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 6 (6)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 6 (6)
Presyncope (Nervous system disorders) | 5 (5) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 6 (6)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Aortic aneurysm (Vascular disorders) | 4 (4) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
Atrioventricular block second degree (Cardiac disorders) | 3 (3) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Colitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Glaucoma (Eye disorders) | 1 (1) | 6 (6)
Localised infection (Infections and infestations) | 3 (3) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (4)
Upper limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Ureterolithiasis (Renal and urinary disorders) | 3 (3) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 4 (4) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 5 (6)
Vitreous haemorrhage (Eye disorders) | 5 (5) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (4)
Aortic valve stenosis (Cardiac disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Embolism arterial (Vascular disorders) | 5 (5) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 5 (5)
Haematoma (Vascular disorders) | 5 (5) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Infected skin ulcer (Infections and infestations) | 5 (5) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 5 (5) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 4 (4)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Staphylococcal infection (Infections and infestations) | 2 (2) | 4 (4)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Abscess limb (Infections and infestations) | 2 (2) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 5 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Bacteraemia (Infections and infestations) | 3 (4) | 2 (2)
Carotid artery occlusion (Nervous system disorders) | 3 (3) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Cystitis (Infections and infestations) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2) | 3 (3)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 5 (5)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 4 (5)
Prostatitis (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 4 (4)
Sudden death (General disorders) | 2 (2) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Vascular stent stenosis (General disorders) | 3 (3) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2)
Arteriosclerosis (Vascular disorders) | 0 (0) | 4 (4)
Atrioventricular block (Cardiac disorders) | 1 (1) | 3 (3)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 3 (3)
Diabetic retinopathy (Eye disorders) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 4 (4) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 3 (3)
Impaired healing (General disorders) | 1 (1) | 3 (4)
Intermittent claudication (Vascular disorders) | 2 (3) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Osteomyelitis acute (Infections and infestations) | 2 (2) | 2 (2)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Peripheral artery thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Wound infection (Infections and infestations) | 1 (1) | 3 (3)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Aortic dissection (Vascular disorders) | 3 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Arterial disorder (Vascular disorders) | 0 (0) | 3 (3)
Arthritis bacterial (Infections and infestations) | 3 (3) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Brain injury (Nervous system disorders) | 3 (3) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 2 (2)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Dementia (Nervous system disorders) | 0 (0) | 3 (3)
Device failure (Product Issues) | 2 (2) | 1 (1)
Diabetic gangrene (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (2) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Epididymitis (Infections and infestations) | 1 (1) | 2 (2)
Facial paralysis (Nervous system disorders) | 1 (1) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Groin abscess (Infections and infestations) | 2 (2) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic enzyme increased (Investigations) | 3 (3) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Hypertensive emergency (Vascular disorders) | 3 (3) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 3 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Liver function test increased (Investigations) | 2 (2) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (5) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 3 (3) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Renal artery stenosis (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 2 (2) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 3 (3)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 2 (2)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Abscess soft tissue (Infections and infestations) | 2 (2) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Cardiac asthma (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cardiomegaly (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 2 (2)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Diabetic vascular disorder (Vascular disorders) | 2 (2) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Essential hypertension (Vascular disorders) | 1 (1) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 2 (2)
Graft infection (Infections and infestations) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
IIIrd nerve paresis (Nervous system disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral discitis (Infections and infestations) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Leriche syndrome (Vascular disorders) | 0 (0) | 2 (2)
Liver abscess (Infections and infestations) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Myelopathy (Nervous system disorders) | 0 (0) | 2 (2)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Osteitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Perirectal abscess (Infections and infestations) | 2 (3) | 0 (0)
Pneumonia viral (Infections and infestations) | 2 (2) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (4) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Venous thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 2 (2)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Accidental death (General disorders) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acoustic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Aortoenteric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Articular calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aspiration bronchial (Investigations) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Basilar artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Biliary ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 1 (1)
Blood ketone body increased (Investigations) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breathing-related sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Brugada syndrome (Cardiac disorders) | 1 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Candiduria (Infections and infestations) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac complication associated with device (General disorders) | 1 (1) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cellulitis gangrenous (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Choroidal detachment (Eye disorders) | 1 (1) | 0 (0)
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Citrobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Citrobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 1 (1) | 0 (0)
Corneoconjunctival intraepithelial neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0)
Coronary no-reflow phenomenon (Cardiac disorders) | 1 (1) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Dengue haemorrhagic fever (Infections and infestations) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Device extrusion (Product Issues) | 1 (1) | 0 (0)
Device issue (Product Issues) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Diabetic mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Emphysematous pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Femoral artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glomerulonephritis acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster infection neurological (Infections and infestations) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypotony of eye (Eye disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
IIIrd nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Impulse-control disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1)
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Kidney contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lymph node fibrosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphorrhoea (Vascular disorders) | 0 (0) | 1 (1)
Lymphostasis (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Mixed dementia (Nervous system disorders) | 0 (0) | 1 (1)
Mononeuritis (Nervous system disorders) | 0 (0) | 1 (1)
Mononeuropathy multiplex (Nervous system disorders) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Necrobiosis (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Nerve degeneration (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuromyopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Normochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Palatal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatic duct stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia moraxella (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Post stroke seizure (Nervous system disorders) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Posterior capsule rupture (Eye disorders) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Prostatic varices (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (2) | 0 (0)
Radial nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectosigmoid cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Retinopathy proliferative (Eye disorders) | 1 (1) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Septic embolus (Infections and infestations) | 1 (1) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue inflammation (General disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord herniation (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternitis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subclavian artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thyroid function test normal (Investigations) | 0 (0) | 1 (1)
Tongue abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Treatment noncompliance (General disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Venous occlusion (Vascular disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Vertebral artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT02465515/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT02465515/SAP_001.pdf